CLINICAL TRIAL: NCT00380354
Title: A Two-centre, Randomised, Double-blind, Placebo-controlled, 2-period Cross-over Study to Evaluate the Effect of Treatment With Repeat Doses of Inhaled GSK256066 on the Allergen-induced Late Asthmatic Response in Subjects With Mild Asthma
Brief Title: Study To Evaluate GSK256066 In Subjects With Mild Bronchial Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPA101985
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Asthma; Mild Asthma
Keywords: allergen; methacholine; GSK256066; mild asthmatics; repeat dose; challenge; late asthmatic response
MeSH Terms: conditions — Asthma | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066

SUMMARY:
This study will evaluate the efficacy and safety of GSK256066 in the treatment of subjects with mild bronchial asthma, using a number of clinical and biological markers of efficacy.

ELIGIBILITY:
Inclusion criteria

* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta -agonist therapy by inhalation.
* Pre-bronchodilator FEV1 >75% of predicted at screening.
* Non-smoker
* Demonstration of a positive reaction to at least one allergen from a battery of allergens (including house dust mite, grass pollen and cat hair on skin prick testing at screening, or within 12 months of study start.
* Have Asthmatic response
* Able and willing to give written informed consent to take part in the study.
* Available to complete all study measurements.

Exclusion criteria:

* History of cardiovascular disease
* Clinically significant abnormalities in safety laboratory analysis at screening including any subject who has greater than "trace urine protein levels" following urinalysis at screening.
* History of hayfever
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
* The subject has tested positive for HIV antibodies.
* The subject has positive drugs of abuse test.
* Subjects weighing less than 50kg are to be excluded from participating in the study.
* The subject has participated in a study with a new molecular entity during the previous 3 months.
* History of being unable to tolerate or complete methacholine, and/or allergen challenge tests.
* There is a risk of non-compliance with study medication or study procedures.
* History of blood donation (450 mL) within 2 months of starting the clinical study.
* The subject regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female. One unit of alcohol is defined as a medium (125 ml) glass of wine, half a pint (250 ml) of beer or one measure (24 ml) of spirits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Asthmatic response | after 7 days of treatment

SECONDARY OUTCOMES:
FEV1 Concentration of exhaled nitric oxide | on day 8 of each treatment period
Incidence of treatment emergent adverse events | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Singh D, Petavy F, Macdonald AJ, Lazaar AL, O'Connor BJ. The inhaled phosphodiesterase 4 inhibitor GSK256066 reduces allergen challenge responses in asthma. Respir Res. 2010 Mar 1;11(1):26. doi: 10.1186/1465-9921-11-26. PMID 20193079